CLINICAL TRIAL: NCT02815085
Title: Pilot to Assess Feasibility of Using RecoverLINK Technology to Supplement Outpatient Care for Heart Failure Patients
Brief Title: RecoverLINK Technology Pilot for HF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RecoverLINK (Industry)
Collaborators: Mount Sinai Hospital, New York (Other); Digital Health Marketplace (previously Pilot Health Tech NYC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IF1793800
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: heart failure; mHealth
MeSH Terms: conditions — Heart Failure

ARMS (1):
- RecoverLINK technology (Experimental): RecoverLINK is a two-part mHealth technology designed to supplement traditional care transitional programs for heart failure (HF) patients.
  Interventions: Other: RecoverLINK technology

INTERVENTIONS:
Other: RecoverLINK technology — HF patients will receive the RecoverLINK app upon study enrollment for 30-days. The Mount Sinai HF care team will interact with patients via the RecoverLINK cloud-based system during this period

SUMMARY:
The primary objective is to examine feasibility of incorporating RecoverLINK into the standard of care as a function of (i) user engagement, (ii) user satisfaction, and (iii) workflow efficiency. As secondary objectives, the investigators will collect preliminary data to examine the association between patient engagement with the RecoverLINK app and (i) changes in patient knowledge and behavior, and (ii) hospital readmission(s) at 30, 60, and 90-day time periods post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure (HF) patients with a rapid follow up appointment scheduled at the Mount Sinai HF clinic
* English-speaking
* With either access to (i) an iOS smart device or (ii) wifi at-home

Exclusion Criteria:

Patients meeting any of the following criteria:

* A heart transplant
* A mechanical circulatory support (MCS) device
* An altered mental status
* Serious co-morbidities (as identified by Mount Sinai team)
* Cognitive impairments (as identified by Mount Sinai team)
* Inability to use technology (as identified by Mount Sinai team)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
User engagement: # symptom surveys completed/30 days | 30 days
User satisfaction: Percent patients report "satisfied" via post-program survey | 30 days
Workflow efficiency: mean/median time to resolution of patient alerts | 30 days

SECONDARY OUTCOMES:
Mean difference in pre/post SCHIFI score | 30 days
Hospital admission | 30, 60, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sean Pinney, MD, Principal Investigator — The Mount Sinai Hospital
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States